CLINICAL TRIAL: NCT02291302
Title: School Inner-City Asthma Intervention Study
Brief Title: School Inner-City Asthma Intervention Study (SICAS-2)
Acronym: SICAS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: U01AI110397 (NIH); U01AI110397 (NIH)
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Environmental Intervention (Active Comparator): Active Classroom air purifiers and school integrated pest management environmental intervention
  Interventions: Other: integrated pest management; Other: air purifier
- Sham and Control (control) (Placebo Comparator): Sham air purifiers and no school integrated pest management environmental intervention
  Interventions: Other: No intervention (control)
- Active Air Purifier and Control (Placebo Comparator): Active air purifiers and no school integrated pest management environmental intervention
  Interventions: Other: air purifier
- Sham and Inegrated Pest (Sham Comparator): Sham air purifiers and active school integrated pest management
  Interventions: Other: integrated pest management

INTERVENTIONS:
Other: integrated pest management — integrated pest management and environmental strategy
  Arms: Environmental Intervention; Sham and Inegrated Pest
Other: air purifier — air purifiers
  Arms: Active Air Purifier and Control; Environmental Intervention
Other: No intervention (control) — no integrated pest management and sham air purifier
  Arms: Sham and Control (control)

SUMMARY:
The investigators goal is to determine the efficacy of school/classroom based environmental intervention in reducing asthma morbidity in urban schoolchildren.

DETAILED DESCRIPTION:
Our proposal builds upon our established, successful school-based infrastructure to determine whether a school/classroom intervention will efficiently and effectively improve asthma morbidity by reducing these exposures. Our goal is to determine the efficacy of school/classroom based environmental intervention in reducing asthma morbidity in urban schoolchildren. Our central hypothesis is that reducing classroom/school exposure to mouse allergen, mold, and particulate pollutants will decrease asthma morbidity in students with asthma. The investigators plan to test this hypothesis in an intervention study of 300 elementary students with asthma from multiple classrooms in inner-city elementary schools. Our clinical trial aims are to determine the effectiveness of a school/classroom based environmental intervention (school integrated pest management and classroom air purifying filter units within these schools) to reduce asthma morbidity. Our mechanistic aim is to test the hypothesis that effects of school/classroom-based environmental interventions on symptoms/other measures of asthma control occur through changes in gene methylation or expression in pathways (and secondarily, in genes) relevant to airway function and asthma. This will expand our understanding of asthma immunopathogenesis and create opportunities to identify potential novel targets for asthma therapy.

ELIGIBILITY:
Inclusion Criteria:

* grades K-8 with asthma attending sampling/intervention schools

Exclusion Criteria:

* moving schools

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD, MS, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ruran HB, Maciag MC, Murphy SE, Phipatanakul W, Hauptman M. Cross-sectional study of urinary biomarkers of environmental tobacco and e-cigarette exposure and asthma morbidity. Ann Allergy Asthma Immunol. 2022 Sep;129(3):378-380. doi: 10.1016/j.anai.2022.06.001. Epub 2022 Jun 7. No abstract available. PMID 35688366
- [Derived] Phipatanakul W, Koutrakis P, Coull BA, Petty CR, Gaffin JM, Sheehan WJ, Lai PS, Bartnikas LM, Kang CM, Wolfson JM, Samnaliev M, Cunningham A, Baxi SN, Permaul P, Hauptman M, Trivedi M, Louisias M, Liang L, Thorne PS, Metwali N, Adamkiewicz G, Israel E, Baccarelli AA, Gold DR; School Inner-City Asthma Intervention study team. Effect of School Integrated Pest Management or Classroom Air Filter Purifiers on Asthma Symptoms in Students With Active Asthma: A Randomized Clinical Trial. JAMA. 2021 Sep 7;326(9):839-850. doi: 10.1001/jama.2021.11559. PMID 34547084
- [Derived] Kantor DB, Petty CR, Phipatanakul W, Gaffin JM. Transcutaneous CO-oximetry differentiates asthma exacerbation and convalescence in children. J Allergy Clin Immunol. 2018 Aug;142(2):676-678.e5. doi: 10.1016/j.jaci.2018.02.048. Epub 2018 Apr 16. No abstract available. PMID 29673798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest
Started | 59 | 59 | 59 | 59
Completed | 59 | 59 | 59 | 59
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest | Total
Number analyzed (Participants) | 59 | 59 | 59 | 59 | 236
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 8.2 (1.9) | 7.9 (1.9) | 8.3 (2.2) | 8.2 (2.0) | 8.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 32 | 33 | 113
  Male | 33 | 37 | 27 | 26 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 35 | 32 | 33 | 138
  Not Hispanic or Latino | 21 | 21 | 25 | 26 | 93
  Unknown or Not Reported | 0 | 3 | 2 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 17 | 12 | 15 | 13 | 57
  White | 21 | 33 | 20 | 26 | 100
  More than one race | 1 | 2 | 8 | 6 | 17
  Unknown or Not Reported | 17 | 11 | 15 | 12 | 55
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 59 | 59 | 236
Maximum Number of Days With Asthma Symptoms Within 2 Weeks [Mean (Standard Deviation); unit: days] | 2.0 (3.2) | 3.0 (4.7) | 1.5 (3.4) | 2.4 (4.2) | 2.2 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Number of Days With Asthma Symptoms Within 2 Weeks
Description: Maximum number of
  1. Days with wheezing, tightness in the chest, or cough and/or
  2. Nights with disturbed sleep as a result of asthma and/or
  3. Days on which the child had to slow down or discontinue play activities because of asthma This is defined as a cumulative assessment from the different variables listed in the Measure Description
Time Frame: up to 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest
Number analyzed (Participants) | 59 | 59 | 59 | 59
days | 2.2 (3.5) | 2.7 (4.4) | 1.2 (2) | 2.1 (3.6)

2. Other Pre Specified Outcome: Lung Function
Description: Spirometry measure of forced expiration volume in 1 second
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of predicted
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest
Number analyzed (Participants) | 55 | 48 | 57 | 46
percentage of predicted | 95.5 (18.5) | 99.2 (16.9) | 97 (14.1) | 94.9 (16.1)

3. Other Pre Specified Outcome: School Absences
Description: Number of school days missed because of asthma/ 2 weeks
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days/2 weeks
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest
Number analyzed (Participants) | 51 | 51 | 54 | 46
days/2 weeks | 0.15 (0.61) | 0.18 (0.75) | 0.16 (0.74) | 0.07 (0.33)

4. Other Pre Specified Outcome: Composite Asthma Severity Index
Description: [a comprehensive severity scale of day symptoms and albuterol use, night symptoms and albuterol use, controller treatment, lung function measures, and exacerbations], health care utilization, and pulmonary function testing (PFT's) including FEV1; FEV1/FVC, FEF25-75. CASI ranges from 0 (lowest) -20 points (highest) with a minimal clinically important difference of 0.49 points. The higher score is worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest
Number analyzed (Participants) | 51 | 51 | 54 | 46
score on a scale | 2.9 (2.2) | 2.8 (2.4) | 3.1 (2.5) | 2.9 (2.2)

5. Post Hoc Outcome: Classroom Viral Exposure
Description: Classroom viral exposure will be assessed using two approaches:
  1. Airborne respiratory viral exposure (copies/m3)
  2. School viral exposure (assessed with virome sequencing)
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-12

6. Post Hoc Outcome: Classroom Microbiome
Description: The classroom microbiome will be assessed with deep metagenomics sequencing
Time Frame: 1 year
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: until study completion an average of 1 year
Arm/Group | Environmental Intervention | Sham and Control (Control) | Active Air Purifier and Control | Sham and Inegrated Pest
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT02291302/Prot_SAP_000.pdf